CLINICAL TRIAL: NCT03423212
Title: Just Do You Program for Young Adults With Serious Mental IIlness: A Randomized Controlled Trial
Brief Title: Just Do You Program for Young Adults With Serious Mental IIlness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R34MH111861-01 (NIH)
Record Dates: First submitted 2018-01-04; First posted 2018-02-06 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2020-09

CONDITIONS: Depression; Bipolar Disorder; Psychosis; Anxiety Disorders
MeSH Terms: conditions — Depression; Bipolar Disorder; Psychotic Disorders; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Condition (Experimental): Participants assigned to the experimental arm will be enrolled in the 2-session Just Do You intervention described elsewhere.
  Interventions: Behavioral: Just Do You
- Treatment as Usual Condition (No Intervention): Participants assigned to treatment as usual will receive the PROS program that is standard in the agencies without any additional intervention.
- Active Control Condition (Active Comparator): Participants assigned to the active control condition will receive the PROS program that is standard in the agencies, and a two-session curriculum on maintaining healthy relationships, which is an identified issue for the population.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Just Do You — Just Do You is an intervention designed to keep young adults connected to their professional behavioral health treatments. It is a brief two-module engagement program that utilizes a hybrid provider team of a licensed clinician and peer to increase young adult engagement in adult outpatient day programs (i.e., New York State Personalized Recovery Oriented Services). The first session consists of the following components: 1) Welcome; Group Guidelines, Purpose, 2) Discuss Recovery Principles; Narrative of Role Model; 3) Video of Celebrity Service User and Discussion, and 4) Recovery Goals (and role of services in that). The second session consists of: 1) What are services & how can they help? 2) Visual art exercise -- Cause of SMI and validation, 3) Maintaining my Medicaid Insurance, and 4) Discussion of Systemic Barriers.
  Arms: Experimental Condition
Behavioral: Active Control — The active control condition will receive the PROS program that is standard in the agencies, and a two-session curriculum on maintaining healthy relationships, which is an identified issue for the population.
  Arms: Active Control Condition

SUMMARY:
Just Do You is a young-adult-centered and theoretically guided intervention that has shown promise for keeping young adults connected to their professional treatments, while also enhancing their hope for the future and their own recovery. Just Do You is a brief two-module engagement program that utilizes a hybrid provider team of a licensed clinician and peer to address mistrust, lack of hope for the future, stigma concerns, literacy and a sense of efficacy early on when young adults begin a new service experience in adult outpatient day programs (i.e., New York State Personalized Recovery Oriented Services). The aim of this study is to test Just Do You through a moderately-sized randomized trial in order to see if it improves initial and secondary engagement among young adults with serious mental health conditions. The program is designed as an orientation to services, coupled with a curriculum designed to enhance motivation and agency, and keep young adults connected to their care.

This study utilizes a randomized controlled trial to test the preliminary impact of the intervention, compared to best available services (treatment as usual, TAU) at two outpatient programs for adults with serious mental illnesses (n = 195). The program was adapted to two-sessions from the piloted four-session version through conversations with leadership at partnering agencies. The intervention involves intensive staff training and 24 months of ongoing provision, monitoring and supervision of the program. Quantitative survey data will be collected at baseline (pre), 2 weeks (post), 1 month, and 3 months. In this intention-to-treat analysis, we will conduct basic omnibus analyses to examine whether Just Do You leads to improved outcomes relative to TAU utilizing t tests across treatment conditions for each outcome measure specified. The investigators will likewise examine whether changes in the proposed mediating variables differ across groups.

DETAILED DESCRIPTION:
Background

Young adults have elevated rates of serious mental illnesses and they often do not receive consistent mental health care. This is a considerable challenge for public health, as most often mental health conditions persist into adulthood. Continuing to engage this population in their professional mental health treatment has been a pervasive challenge globally. Few mental health interventions have been designed specifically for young adults and none are conceptualized as meta-interventions or orientation programs. Just Do You is a young-adult-centered and theoretically guided intervention that has shown promise for keeping young adults connected to their professional treatments, while also enhancing their hope for the future and their own recovery. Just Do You is a brief two-module engagement program that utilizes a hybrid provider team of a licensed clinician and peer to address mistrust, lack of hope for the future, stigma concerns, literacy and a sense of efficacy early on when young adults begin a new service experience in adult outpatient day programs (i.e., New York State Personalized Recovery Oriented Services).

Methods/design

This study utilizes a randomized controlled trial to test the preliminary impact of the intervention, compared to best available services (treatment as usual, TAU) at two outpatient programs for adults with serious mental illnesses (n = 195). The program was adapted to two-sessions from the piloted four-session version through conversations with leadership at partnering agencies. The intervention involves intensive staff training and 24 months of ongoing provision, monitoring and supervision of the program. Quantitative survey data will be collected at baseline (pre), 2 weeks (post), 1 month, and 3 months. In this intention-to-treat analysis, the investigators will conduct basic omnibus analyses to examine whether Just Do You leads to improved outcomes relative to TAU utilizing t tests across treatment conditions for each outcome measure specified. The investigators will likewise examine whether changes in the proposed mediating variables differ across groups.

Discussion

The aim of this study is to test Just Do You through a moderately-sized randomized trial in order to see if it improves initial and secondary engagement among young adults with serious mental health conditions. The program is designed as an orientation to services, coupled with a curriculum designed to enhance motivation and agency, and keep young adults connected to their care. Continuity of care among this population is a serious challenge and Just Do You has the potential to address this challenge in the service system for poor, young adults living in low-resourced communities. If it is shown to be successful in this setting, it could likely be used to address the continuity of care issue more broadly in additional settings that serve young adults with serious mental illness. It may enhance the menu of care options for those who have been recently diagnosed with a serious mental health condition, providing them with an orientation for how professional mental health care can help them. The program is recovery-oriented, builds on the best evidence to date, and is in line with both local and national health care reform efforts.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 28
* living with a serious mental illness (i.e., mood, anxiety, schizophrenia-spectrum)
* attending personalized recovery-oriented services (PROS)
* formerly involved with public systems of care

Exclusion Criteria:

* cognitive impairments (i.e., young adult cannot understand consent process or IQ<70)
* non-English speaking (we will include individuals whose primary language is not English, but are able to comprehend and speak English).

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-03-07 (Actual); Study Completion 2020-03-07 (Actual)

PRIMARY OUTCOMES:
Adherence to PROS program | Assessed 4 weeks following baseline
  Past week attendance to mental health appointments at PROS
Adherence to PROS program | Assessed 3 months following baseline
  Past week attendance to mental health appointments at PROS

SECONDARY OUTCOMES:
Adherence to medication | Assessed 4 weeks following baseline
  Past week adherence to mental health-related medications
Adherence to medication | Assessed 3 months following baseline
  Past week adherence to mental health-related medications
Client Engagement in Child Protective Services Scale | Assessed 4 weeks following baseline
  This scale is altered to measure young adult engagement in PROS services. The scale includes 8 questions and responses will be summed. The range for the scale is 8 to 40, with higher scores indicating higher levels of engagement.
Client Engagement in Child Protective Services Scale | Assessed 3 months following baseline
  This scale is altered to measure young adult engagement in PROS services. The scale includes 8 questions and responses will be summed. The range for the scale is 8 to 40, with higher scores indicating higher levels of engagement.

OTHER OUTCOMES:
Center for Epidemiological Studies Depression Scale | Assessed 3 months following baseline
  This is a standardized measure of depression. The range on the scale is 0 to 60. Scores will be summed. Higher scores indicated higher levels of depression.
Global Measure of Perceived Stress | Assessed 4 weeks following baseline
  This is a standardized measure of recent stress. The range on the scale is 0 to 56. Scores will be summed. Higher scores indicated higher levels of stress.
Inventory of Attitudes Toward Seeking Mental Health Services | Assessed 4 weeks following baseline
  The investigators will use the stigma subscale of the Inventory of Attitudes Toward Seeking Mental Health Services. The range of the measure is 0 to 48, with higher scores indicating higher levels of stigma. For this study the score will be summed.
Inventory of Attitudes Toward Seeking Mental Health Services | Assessed 3 months following baseline
  The investigators will use the stigma subscale of the Inventory of Attitudes Toward Seeking Mental Health Services. The range of the measure is 0 to 48, with higher scores indicating higher levels of stigma. For this study the score will be summed.
Group-Based Medical Mistrust Scale | Assessed 4 weeks following baseline
  Standardized measure of mistrust of mental health services. The range for the measure is 4 to 20. For this study the scores will be summed, with higher scores indicating more mistrust.
Group-Based Medical Mistrust Scale | Assessed 3 months following baseline
  Standardized measure of mistrust of mental health services. The range for the measure is 4 to 20. For this study the scores will be summed, with higher scores indicating more mistrust.
The Hope Scale | Assessed 4 weeks following baseline
  This is a standardized measure of hope. The scores will be summed. The range is 8 to 96, with higher scores indicating higher levels of hope.
The Hope Scale | Assessed 3 months following baseline
  This is a standardized measure of hope. The scores will be summed. The range is 8 to 96, with higher scores indicating higher levels of hope.
Self-Efficacy/Advocacy | Assessed 4 weeks following baseline
  Perceived Behavioral Control (4-items adapted from autonomy factor and 3-items from capacity factor). The scores will be summed. For the autonomy factor, the range is 4 to 16, with higher scores indicating more control and autonomy. For the capacity factor, the range is 3 to 12, with higher scores indicating less capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle R Munson, PhD, Principal Investigator — New York University; James Jaccard, PhD, Principal Investigator — New York University
Locations (1):
- Mt Eden Personalized Recovery Oriented Services, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munson MR, Jaccard J, Scott LD Jr, Moore KL, Narendorf SC, Cole AR, Shimizu R, Rodwin AH, Jenefsky N, Davis M, Gilmer T. Outcomes of a Metaintervention to Improve Treatment Engagement Among Young Adults With Serious Mental Illnesses: Application of a Pilot Randomized Explanatory Design. J Adolesc Health. 2021 Nov;69(5):790-796. doi: 10.1016/j.jadohealth.2021.04.023. Epub 2021 Jun 4. PMID 34099390
- [Derived] Munson MR, Jaccard JJ, Scott LD Jr, Narendorf SC, Moore KL, Jenefsky N, Cole A, Davis M, Gilmer T, Shimizu R, Pleines K, Cooper K, Rodwin AH, Hylek L, Amaro A. Engagement intervention versus treatment as usual for young adults with serious mental illness: a randomized pilot trial. Pilot Feasibility Stud. 2020 Jul 23;6:107. doi: 10.1186/s40814-020-00650-w. eCollection 2020. PMID 32714561

DOCUMENTS (1):
  • Informed Consent Form (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT03423212/ICF_000.pdf